CLINICAL TRIAL: NCT01879046
Title: Regenerative Medicine of Articular Cartilage: Characterization and Comparison of Chondrogenic Potential and Immunomodulatory Adult Mesenchymal Stem Cells
Acronym: ARTHROSTEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC12_0394
Record Dates: First submitted 2013-05-27; First posted 2013-06-17 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Knee Osteoarthritis
Keywords: Mesenchymal stem cells; articular cartilage; tissue engineering; immunomodulation; osteo-arthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical intervention (Experimental): Blood, bone marrow and Hoffa's fat pad samplings during surgical intervention
  Interventions: Procedure: arthroplasty

INTERVENTIONS:
Procedure: arthroplasty — Blood, bone marrow, synovial fluid and Hoffa's fat pad samplings

SUMMARY:
Articular cartilage can be the seat of many diseases including osteoarthritis and traumatic defaults. The cartilage has no intrinsic ability to repair resulting at long term in function loss in the joints. Currently available treatments are not satisfactory in the long term, the use of mesenchymal stem cells appears to be promising due to their ability to multipotency and immunomodulation properties. This project aims to determine the most appropriate source for regenerative medicine of cartilage stem cells from tissue taken during arthroplasty in patients with osteoarthritis. These cells will be tested for different chondrogenic markers. The success of this project will consider the implementation of a strategy for regenerative medicine in bone and joint diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Patients with knee osteoarthritis
* Patients requiring total knee arthroplasty
* Patients who signed the consent form

Exclusion Criteria:

* Patients aged less than 18 years
* Major Patients under guardianship
* Pregnant woman
* Infectious pathology or progressive tumor
* Refusal to participate in the study
* State of immunosuppression
* Congenital or acquired malformation resulting in a deformation of the knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Increased expression of chondrogenic markers | up to 3 years
  Increased expression of chondrogenic markers will be Evaluated by different techniques:
  in vitro: Histology fit for chondrogenic markers, RT-PCR on the following markers aggrecan, type II collagen, Sox9, Comp, type IX collagen
  in vivo: In a second step, differentiated MSCs are implanted in vivo after combination with a hydrogel subcutaneously in nude mice. The formation of a neo cartilage tissue will be assessed by histology for type II collagen and aggrecan

SECONDARY OUTCOMES:
Increasing secretion of anti-inflammatory molecules in vitro | up to 3 years
  Increasing secretion of anti-inflammatory molecules in vitro will be tested by several techniques:
  Microfluidic cards (TLDA assays) for the analysis of the expression of genes involved in inflammation and in the secretion of anti-inflammatory molecules Inhibition of proliferation of autologous T cells activated or not Assay for anti-inflammatory and pro-inflammatory molecules Analysis of the expression of surface markers by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ronan Guillou, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France